CLINICAL TRIAL: NCT04036734
Title: Does Longitudinal or Transverse Orientation of Ultrasound Probe Improve Cannulation Success in Minimally Invasive Venous Surgery. A Randomized Controlled Trial.
Brief Title: Longitudinal or Transverse Orientation of Ultrasound Probe in Minimally Invasive Venous Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Thomas Aherne, Research Fellow Vascular Surgery, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USGSV
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Varicose Veins; Endovenous Procedures; Venous Access
MeSH Terms: conditions — Varicose Veins | interventions — Global Longitudinal Strain

STUDY DESIGN:
Intervention Model Description: Parallell block randomised groups
Who Masked: Participant
Masking Description: Intraoperative draping to obscure patient view
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverse Ultrasound Orientation (Active Comparator): Transverse placement of ultrasound to long axis of target lower limb vein
  Interventions: Diagnostic Test: Transverse
- Longitudinal Ultrasound Orientation (Experimental): Longitudinal placement of ultrasound to long axis of target lower limb vein
  Interventions: Diagnostic Test: Longitudinal

INTERVENTIONS:
Diagnostic Test: Longitudinal — Longitudinal orientation of ultrasound to long axis of vein to guide access needle
  Arms: Longitudinal Ultrasound Orientation
Diagnostic Test: Transverse — Transverse orientation of ultrasound to long axis of vein to guide access needle
  Arms: Transverse Ultrasound Orientation

SUMMARY:
Longitudinal ultrasound orientation during central venous cannulation has been suggested by a number of radomised studies to offer superior cannulation rates. This technique may offer a simple, safe and cost-neutral step to improve cannulation rates in the widely performed minimally invasive endovenous intervention.

DETAILED DESCRIPTION:
Varicose veins are an extremely common disorder and negatively impact on patient quality of life. In recent years minimally invasive venous treatments for varicose veins (MIVT) have emerged as an effective alternative to open surgery. It is associated with a reduction in peri-operative morbidity, recovery time and increased quality of life scores when compared with open surgical stripping4. Furthermore, MIVT is now widely carried out under local anaesthesia.

Typically, MIVT requires cannulation, under ultrasound guidance, of either the great or small saphenous vein in the lower extremity to allow subsequent passage of a venous catheter. This cannulation technique is widely used for venous and arterial cannulation throughout the body. It entails utilising an ultrasound probe in either a longitudinal or transverse orientation (to the target vein) to guide an entry needle into a target vessel. The longitudinal orientation, while unstable, offers better visualisation of the vein when performed accurately. Conversely, the transverse approach is very stable with poorer visualisation of the target vessel. As such, no definitve guidance is available to guide treating physicians as to the optimal orientation with a wide variation among practitioners.

The cannulation process for MIVT is often further challenged by both the small calibre and tendency toward vasospasm of target veins. Failure of cannulation may result in greater rates of conversion to open surgery exposing the patient to the the higher rate of morbidity associated with open surgery. More importantly, repeated cannulation results in significant discomfort and hence a reduction in patient satisfaction.

Longitudinal ultrasound orientation during venous cannulation has been suggested by a number of radomised studies to offer superior cannulation rates of cannulation. This technique may offer a simple, safe and cost-neutral step to improve cannulation rates in the widely performed MIVT.

The authors propose a blinded randomized controlled study to investigate the effects of ultrasound orietation on cannulation rates in MIVT. To test this hypothesis we plan to randomise 100 patients undergoing MIVT to either venous cannulation with transverse or longitudinal orientation of the ultrasound probe.

ELIGIBILITY:
Inclusion Criteria:

* For minimally invasive venous surgery of the lower limb (Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification score 2 of greater)
* Intervention requiring venous cannulation of axial lower limb vein
* Full consent
* >18 years
* No concomitant deep venous incompetence

Exclusion Criteria:

* General anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Overall successful Cannulation rate as a percentage | Immediate
  Overall successful cannulation of the target axial lower limb vein for endovenous treatment. Successful cannulation will be defined as intraluminal placement of the access cannula in the targeted axial vein.

SECONDARY OUTCOMES:
Time in seconds to cannulation | Immediate
  Time from skin puncture to successful placement of access catheter in the target vein
Number of cannulation attempts | Immediate
  Number of times the skin is pierced in an attempt to cannulate the target vein
Peri-cannulation pain | Immediate
  Pain will be measured using a visual analogue scale of 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Stewart R Walsh, Principal Investigator — National University of Ireland, Galway
Locations (1):
- Saolta University Hospital Group, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT04036734/Prot_000.pdf